CLINICAL TRIAL: NCT06187181
Title: Hyoid Displacement During Swallowing Function for Completely Edentulous Subjects Rehabilitated With Mandibular Implant Retained Overdenture
Brief Title: Hyoid Displacement During Swallowing Function for Completely Edentulous Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A19061222
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-12

CONDITIONS: Prosthesis Durability
Keywords: Hyoid bone.; implant.; overdenture; swallowing.
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G. I : Completely edentulous patients (Placebo Comparator): videofluroscopy for completely edentulous patients
  Interventions: Radiation: videofluroscopy
- G.II: patients with complete dentures (Active Comparator): complete denture construction for edentulous patient and videofluroscopy evaluation
  Interventions: Procedure: implant overdenture; Radiation: videofluroscopy
- G.III: patients with implant overdentures (Active Comparator): construction of implant overdenture and videofluroscopy evaluation
  Interventions: Procedure: implant overdenture; Radiation: videofluroscopy

INTERVENTIONS:
Procedure: implant overdenture — . Videofluoroscopy swallowing evaluation was done using 10 ml of thin liquid bolus at three different oral conditions: Without dentures (WOD), with the conventional complete denture (CDs) and with mandibular implant retained overdenture (IODs).
  Arms: G.II: patients with complete dentures; G.III: patients with implant overdentures
Radiation: videofluroscopy — videofluroscopy evaluation of swallowing function

SUMMARY:
To investigate the effect of wearing mandibular implant retained overdentures on superior and anterior hyoid displacement during swallowing process.

DETAILED DESCRIPTION:
New conventional complete denture with optimal flange extension and well established lingualized balanced occlusal scheme was constructed for every patient. To construct the radiographic stent, clear acrylic resin duplicate for the mandibular denture was constructed, several small holes were made on the polished surface of the duplicate. These holes were filled with radio-opaque gutta-percha points to act as a reference points during determination of the quantity of available bone for implant placement and for construction of stereolithographic surgical guide.

Cone beam computerized tomography [i-CAT] was used to construct the stereolithographic surgical guide by applying dual scan technique. By using the surgical guide, two dental implants (Dentium implants, 12-14mm in length, 3.6-4mm in diameter, Superline II) were placed in the canine regions of the mandibular arch with guided surgical protocol. The patients were instructed to take prophylactic antibiotic two times a day (875mg Amoxicillin and 125mg Clavulanic acid) 24 hours before the surgery and continue after the surgery for seven days. Non-steroidal anti-inflammatory drug was used to control the pain.

After surgery, the complete denture was withdrawn, and the patient was instructed to eat soft diet. After one week, the mandibular denture was relieved and relined with Cold- curing silicon based relining material (Softliner, PROMEDICA). The dentures were delivered to the patients and follow up visits were scheduled. After three to four months, the dental implants were exposed, and the healing abutments were secured to the dental implants. After healing of the soft tissue (7-10 days), the healing abutments were removed, and ball attachments (Dentium ball abutment, Superline II) were screwed to the dental implants. Direct pick-up technique was used to incorporate the housing of the attachments into the fitting surface of the mandibular denture using self-cured acrylic resin material. The occlusion of the overdenture was evaluated to eliminate any premature occlusal contact then the overdenture was delivered to the patient.

Videofluroscopic swallowing study (VFSS):

All subjects were examined by using videofluroscopic swallowing study to evaluate bolus movements. This evaluation was done at three different oral conditions, without complete denture (WCD), after 2 months of conventional complete dentures insertion (CDs), and after 2 months of implant overdenture insertion (IODs). Each patient was instructed to swallow 10 ml of thin liquid {20% barium sulfate (Prontobario H.D®) and 80% water} three times. The records of the videofluroscopic swallowing evaluation were saved to the computer for later analysis. A software Program (EO Program) was used to placing timing on the frame of the video (1/100 second) and analyze the recording by frame by frame data analysis.

a- Spatial measurements: Superior hyoid displacement (vertical movement) and anterior hyoid displacement (horizontal movement) were measured according to dynamic swallowing study performed by Rebecca Leonard & Katherine Kendall during pseudo rest position and during maximum overall hyoid displacement .24 Aline was drawn from anterior superior point of cervical spine 4 (p1) contacting anterior inferior point of cervical spine 2 (p2) and extended superiorly as necessary, then another line was extended from the anterior, inferior portion of the hyoid bone to meet the P1-P2 line at 90-degree intersection. The Measurement from the P1 to the intersection point (Hsup-rest) and from hyoid bone to the intersection point (Hant-rest) were recorded then the video was advanced until the hyoid bone showed maximum overall displacement and the previous procedure was repeated. The measurements from P1 to the intersection point (Hsup-max) and from the hyoid bone to the intersection point (Hant- max) were recoded. The difference between the maximum hyoid position (Hsup-max) and the pseudo rest position (Hsup-rest) in the vertical direction was called the superior hyoid displacement, while the difference between maximum hyoid position (Hant-max) and pseudo rest position (Hant-rest) in the horizontal direction was called anterior hyoid displacements.

B- Temporal measurements:

1. Duration of hyoid maximum elevation (DOHME):

   Measured from the first frame showing maximum hyoid elevation to last frame showing maximum hyoid elevation.
2. Duration of hyoid maximum anterior excursion (DOHMAE):

Measured from the first frame showing maximum anterior hyoid movement to last frame showing maximum anterior hyoid movement.

C- Penetration / aspiration scale:

Penetration was defined as the food bolus enter the airway down to the vocal folds, while aspiration defined as the food bolus enter the airway below the level of the vocal folds.

0= No penetration or aspiration

1. Penetration
2. Aspiration

ELIGIBILITY:
Inclusion Criteria:

* free from any medical problems that may affect the osseointegration of the dental implants
* class I maxillomandibular relationship and free from any previous swallowing problems

Exclusion Criteria:

* participants with temporomandibular joint disorder,
* head and neck surgery,
* sleep apnea
* skeletal deformity

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
swallowing evaluation | after 3 months of denture or overdenture insertion
  hyoid bone displacement evaluation by videofluriscopy

CONTACTS AND LOCATIONS:
Overall Officials: abdallah Ibrahim, PhD, Principal Investigator — Mansoura university, Faculty of dentistry, prosthodontics department
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kern JS, Kern T, Wolfart S, Heussen N. A systematic review and meta-analysis of removable and fixed implant-supported prostheses in edentulous jaws: post-loading implant loss. Clin Oral Implants Res. 2016 Feb;27(2):174-95. doi: 10.1111/clr.12531. Epub 2015 Feb 9. PMID 25664612
- [Derived] Ibrahim AM, Elgamal M, Abdel-Khalek EA. Hyoid displacement during swallowing function for completely edentulous subjects rehabilitated with mandibular implant retained overdenture. BMC Oral Health. 2024 Aug 8;24(1):914. doi: 10.1186/s12903-024-04616-9. PMID 39118020